CLINICAL TRIAL: NCT04550195
Title: A Double-Blind, Placebo-Controlled, Randomized, Single and Multiple Ascending Dose Study of the Safety and Tolerability, and Pharmacokinetics (Including Food Effect, pH Effect and Japanese Bridging Study) of BMS-986337 Following Oral Administration in Healthy Participants
Brief Title: A Study to Evaluate the Safety, Tolerability, and Drug Levels of BMS-986337 When Taken by Mouth by Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IM037-009; 2019-004518-32 (EudraCT Number)
Record Dates: First submitted 2020-09-11; First posted 2020-09-16 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Healthy Volunteers
Keywords: Healthy volunteers
MeSH Terms: interventions — Famotidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (13):
- Part A Single Ascending Dose (SAD) Cohort A1 (Experimental)
  Interventions: Drug: BMS-986337; Other: BMS-986337 Placebo
- Part A SAD Cohort A2 (Experimental)
  Interventions: Drug: BMS-986337; Other: BMS-986337 Placebo
- Part A SAD Cohort A3 (Experimental)
  Interventions: Drug: BMS-986337; Other: BMS-986337 Placebo
- Part A SAD Cohort A4 (Experimental)
  Interventions: Drug: BMS-986337; Other: BMS-986337 Placebo
- Part A SAD Cohort A5 (Experimental)
  Interventions: Drug: BMS-986337; Other: BMS-986337 Placebo
- Part A SAD Cohort A6 (Experimental)
  Interventions: Drug: BMS-986337; Biological: Famotidine
- Part B Multiple Ascending Dose (MAD) Cohort B1 (Experimental)
  Interventions: Drug: BMS-986337; Other: BMS-986337 Placebo
- Part B MAD Cohort B2 (Experimental)
  Interventions: Drug: BMS-986337; Other: BMS-986337 Placebo
- Part B MAD Cohort B3 (Experimental)
  Interventions: Drug: BMS-986337; Other: BMS-986337 Placebo
- Part B MAD Cohort B4 (Experimental)
  Interventions: Drug: BMS-986337; Other: BMS-986337 Placebo
- Part C MAD in Japanese Healthy participants Cohort C1 (Experimental)
  Interventions: Drug: BMS-986337; Other: BMS-986337 Placebo
- Part C MAD in Japanese Healthy participants Cohort C2 (Experimental)
  Interventions: Drug: BMS-986337; Other: BMS-986337 Placebo
- Part C MAD in Japanese Healthy participants Cohort C3 (Experimental)
  Interventions: Drug: BMS-986337; Other: BMS-986337 Placebo

INTERVENTIONS:
Drug: BMS-986337 — Specified Dose on Specified Days
Other: BMS-986337 Placebo — Specified Dose on Specified Days
  Arms: Part A SAD Cohort A2; Part A SAD Cohort A3; Part A SAD Cohort A4; Part A SAD Cohort A5; Part A Single Ascending Dose (SAD) Cohort A1; Part B MAD Cohort B2; Part B MAD Cohort B3; Part B MAD Cohort B4; Part B Multiple Ascending Dose (MAD) Cohort B1; Part C MAD in Japanese Healthy participants Cohort C1; Part C MAD in Japanese Healthy participants Cohort C2; Part C MAD in Japanese Healthy participants Cohort C3
Biological: Famotidine — Specified Dose on Specified Days
  Arms: Part A SAD Cohort A6

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and drug levels of BMS-986337 in healthy participants and in healthy Japanese participants.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant deviation from normal in medical history, physical examination, electrocardiograms (ECGs), and clinical laboratory determinations
* For Japanese cohorts in Part C, must be first-generation Japanese (born in Japan, not living outside of Japan for more than 10 years, and both parents are ethnically Japanese)
* Body mass index (BMI) of 18.0 kg/m^2 to 30.0 kg/m^2, inclusive, at screening; BMI = weight (kg)/height (m)^2
* Women and men must agree to follow specific methods of contraception, if applicable

Exclusion Criteria:

* Women who are of childbearing potential
* Women who are breastfeeding
* Prior exposure to BMS-986278
* Positive nasopharyngeal reverse transcriptase polymerase chain reaction (RT-PCR) test for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) on Day -2

Other protocol-defined inclusion/exclusion criteria apply

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-09-17 (Actual); Primary Completion 2021-03-03 (Actual); Study Completion 2021-03-03 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) | Up to 30 days
Incidence of Serious Adverse Events (SAEs) | Up to 81 days
Incidence of AEs leading to discontinuation | Up to 30 days
Number of clinically significant changes in clinical laboratory values: Hematology tests | Up to 51 days
Number of clinically significant changes in clinical laboratory values: Urinalysis tests | Up to 51 days
Number of clinically significant changes in clinical laboratory values: Clinical chemistry tests | Up to 51 days
Number of clinically significant changes from baseline in vital signs: Heart Rate | Up to 51 days
Number of clinically significant changes from baseline in vital signs: Body Temperature | Up to 51 days
Number of clinically significant changes from baseline in vital signs: Blood Pressure | Up to 51 days
Number of clinically significant changes from baseline in vital signs: Respiratory Rate | Up to 51 days
Number of clinically significant changes in electrocardiogram (ECG) parameters: Heart rate (HR) | Up to 51 days
Number of clinically significant changes from baseline in physical examinations | Up to 51 days
Number of clinically significant changes in ECG parameters: PR interval | Up to 51 days
  PR interval is the time from the onset of the P wave to the start of the QRS complex
Number of clinically significant changes in ECG parameters: QRS duration | Up to 51 days
  QRS can be defined as the electrical impulse as it spreads through the ventricles, indicating ventricular depolarization
Number of clinically significant changes in ECG parameters: QTc-interval (Fridericia's) | Up to 51 days
  QTcF = Corrected QT interval using the Fridericia formula. QT interval is the time from the start of the Q wave to the end of the T wave.
Number of clinically significant changes in ECG parameters: QT interval | Up to 51 days
  The QT interval is the time from the start of the Q wave to the end of the T wave.

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- ICON Plc (PRA Health Sciences) - Netherlands, Groningen, Netherlands

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm